CLINICAL TRIAL: NCT00164892
Title: Selective COX-II Inhibitor as an Adjuvant Therapy in Patients With Resectable Advanced Stomach Cancer ( Histological Staging ≥ T2N1) - A Multi-Centre Prospective Randomised Controlled Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE-2001.463-T
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-11-17 (Estimated); Status verified 2005-09

CONDITIONS: Cancer of Stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — rofecoxib

INTERVENTIONS:
Drug: Oral Vioxx (Rofecoxib)

SUMMARY:
The purpose of this study is to investigate the efficacy of selective COX-II inhibitor in patients with curative resection performed for locally advanced stomach cancer.

DETAILED DESCRIPTION:
Cyclo-oxygenase (COX) is a family of enzymes regulating the conversion of arachidonic acid to prostaglandins. COX-II is an inducible enzyme, which may be upregulated when there are stimuli such as inflammation or hypergastrinaemia. Despite radical surgery, patients with stomach cancer of advanced stages often have a poor prognosis. Reported survival in those with diseases of stage IIIa or above is less than 40%. Methods to improve patients outcome have been explored for decades with little success. In the light of current understanding on the relation between COX-II and stomach cancer, selective COX-II inhibitor may be used as a novel adjuvant therapy after gastrectomy to prevent recurrence of gastric carcinoma. The advantages of COX-II inhibitors are being relatively non-toxic with minimal side effect.

ELIGIBILITY:
Inclusion Criteria:

* Resectable advanced stomach cancer (Tumour stage ≥ T2N1 according to the 5th edition of UICC staging system) without peritoneal or distant metastases.
* Normal renal function

Exclusion Criteria:

* Solid organ metastases
* Poor performance status
* Already on long-term aspirin or NSAID
* Renal or hepatic dysfunction
* Bleeding disorder
* Hypersensitive to COX-II inhibitors/aspirin/NSAID
* No history of myocardial infarct or stoke

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214
Dates: Start 2004-10

PRIMARY OUTCOMES:
Recurrence free survival and the quality of life score within the two years of study period

SECONDARY OUTCOMES:
Overall survival in long term

CONTACTS AND LOCATIONS:
Overall Officials: Enders K.W. Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Combine Gastro-intestinal Cancer Clinic, Hong Kong, China